CLINICAL TRIAL: NCT03451383
Title: Older Breast Cancer Patients: Risk for Cognitive Decline. The Thinking and Living With Cancer (TLC) Study
Brief Title: Older Breast Cancer Patients: Risk for Cognitive Decline
Acronym: TLC
Status: Recruiting | Type: Observational
Sponsor: Georgetown University (Other)
Collaborators: Memorial Sloan Kettering Cancer Center (Other); Indiana University (Other); H. Lee Moffitt Cancer Center and Research Institute (Other); City of Hope Medical Center (Other); Hackensack Meridian Health (Other)
Responsible Party: Principal Investigator, Jeanne Mandelblatt, Professor, Georgetown University
Other Study IDs: 2008-363
Record Dates: First submitted 2018-01-29; First posted 2018-03-01 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Cancer, Breast; Age-related Cognitive Decline; Cognitive Decline
Keywords: breast cancer; cognitive decline
MeSH Terms: conditions — Breast Neoplasms; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A total of up to 27ml of blood will be collected at each time point for APOE and COMT DNA testing, inflammatory biomarkers, plasma AD-pathology markers (Aβ1- 42, tau, p-tau, and neurofilament light chain [NFL]), the receptor for advanced glycation end- products (RAGE) and danger-associated molecular patterns (DAMPs: Aβ, S100 proteins, and HMBG1) and for storage of DNA and RNA for future research. If the subject is unable to provide a blood sample at their visit, 2ml of saliva will be collected using Oragene DNA Collection kits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Breast Cancer Case: Women age 60+ with a newly diagnosed breast adenocarcinoma staged 0-3.
- Non-Cancer Controls: Women age 60+ with no diagnosis of breast cancer.

SUMMARY:
The goal of this study is to evaluate the impact of systemic therapy on cognition in older breast cancer patients, explore change in APE, LM and Cognition domains, measure associations between cognitive decline and QOL, and describe how genetic polymorphisms, inflammatory biomarkers, sleep and physical measures moderate cognitive outcomes. This study is being done nationally, with recruiting sites at Georgetown University, Montgomery General Hospital, Virginia Cancer Specialists, Washington Hospital Center, Reston Breast Care Specialists, Memorial Sloan-Kettering, Moffitt Cancer Center, City of Hope National Medical Center, Hackensack University Medical Center, Indiana University and University of California, Los Angeles.

DETAILED DESCRIPTION:
Cancer is the leading cause of death in the US and breast cancer is the second most common cancer among women in our country. Older women (women 60 and older) presently account for nearly half of all new cases of breast cancer. With the "graying of America" and advances in treatment for breast cancer, the absolute number of older women undergoing breast cancer treatment and surviving their disease will almost double by the year 2030. Systemic hormonal and non-hormonal chemotherapy is credited with improvements in survival, and rates of use of these modalities have increased substantially over the past two decades. Preliminary work has found that older women are interested in chemotherapy even for small returns in survival extension. However, cognitive impairment has been demonstrated in most studies of breast cancer systemic treatments, but virtually all of this research has been conducted in younger populations. Since aging itself is associated with cognitive declines, it seems very likely that older women are particularly vulnerable to the adverse cognitive effects of systemic therapy; our preliminary work strongly suggests that this is the case, but this has never been empirically tested.

This study will be the first large-scale, prospective, controlled investigation to evaluate cognitive changes in older cancer patients and it will provide the basis for the next generation of mechanistic, treatment and intervention studies. These will be important since data from younger patients cannot be directly translated into the older population. Investigators will use the vulnerability model of cancer survivorship to prospectively describe the magnitude of systemic therapy effects on cognition in older (age >60 years) breast cancer patients over a 60 month period, explore change in APE, LM and Cognition domains, test associations between cognition and quality of life (QOL), and evaluate whether genetic polymorphisms, inflammatory biomarkers, sleep and physical measures moderate cognitive outcomes.

To achieve these objectives, investigators have assembled a multi-disciplinary team of oncologists, geriatricians, neurologists, neuro- and cognitive psychologists, behavioral scientists and consumers from Lombardi Comprehensive Cancer Center (LCCC), Memorial Sloan-Kettering Cancer Center (MSKCC), Moffitt Cancer Center, City of Hope National Medical Center (COH), Hackensack University Medical Center (HUMC), Indiana University (IU), Boston University (BU), University of California (UCLA), University of South Florida (USF) and their satellites, will work together to prospectively enroll 850 newly diagnosed older breast cancer cases from LCCC, MSKCC, Moffitt, COH, HUMC, IU and tertiary referral centers with high volumes. An equal number of non-cancer friend controls will be recruited. Friend controls were chosen since they will be similar to patients in most ways except for exposure to cancer and its treatments and they should be motivated to participate. If friends are not available, controls matched to cases on age, education, race, and area (DC/NY/FL/CA/NJ/IU) will be recruited from the community.

Investigators will administer baseline neuropsychological testing prior to any systemic treatment (or at enrollment for controls), survey women about subjective cognitive function, sleep, psychosocial factors, QOL and activities of daily living (IADLS). Subjects will take part in physical measurements, including grip strength, sit to stand and walk speed tests. Investigators will abstract clinical data from medical records. Investigators will obtain blood or saliva to test for APOE, COMT and other genetic polymorphisms at enrollment; these results will not be provided to participants since this is considered a research test). Subjects have the option to provide blood for biomarker research and for biobanking. Subjects will also provide one week of sleep monitoring. Subjects at IU will have the option to participate in neuroimaging. Investigators conduct follow-up interviews and repeat the neuropsychological testing, physical measures, blood/saliva collection, sleep monitoring and optional neuroimaging 12 months after baseline assessment; this time point corresponds to 3-6 months post-treatment among women who receive chemotherapy. Our primary cognitive outcome will be change in summary score on tests in the Attention, Processing Speed, and Executive Function domain, Learning and Memory domain, and Subjective Cognition domain. In secondary analyses, investigators examine changes in scores on additional domains to assess broader cognitive function and examine questions of differential impact.

Data from this study will guide future interventions to better select older women for whom the benefits of systemic therapy outweigh the harms and to develop approaches to mitigate negative consequences of systemic treatment when it is indicated, improving the quality of care for the growing population of older breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

For cancer patients, eligibility includes:

* being female
* Age 60+ at diagnosis of a new primary histological confirmed adenocarcinoma breast cancer
* AJCC stages 0-3 or planning neoadjuvant therapy
* In the judgment of the consenting professional, able to communicate well enough in English through verbal and written communication to complete the study assessments and provide informed consent
* If currently taking psychoactive medications (including, but not limited to anticonvulsants, antidepressants, and anxiolytics), dose must have been stable at least two months prior to enrollment.
* Participant report of no previous or current chemotherapy or hormonal treatment use (anastrazole, exemestane, etc.) This does not include hormonal replacement therapy, synthetic thyroid hormones, etc.

For controls, eligibility includes:

* being female
* Age 60+
* In the judgment of the consenting professional, able to communicate well enough in English through verbal and written communication to complete the study assessments and provide informed consent
* If currently taking psychoactive medications (including, but not limited to anticonvulsants, antidepressants, and anxiolytics), dose must have been stable at least two months prior to enrollment.

Exclusion:

We apply the same exclusion criteria for patients and controls.

* Participant report of a history of formal diagnosis of neurological problems (i.e. Alzheimer's disease, Parkinson's disease, Multiple Sclerosis, Dementia, Seizure Disorders, brain tumors, etc.)
* Participant report of surgery on the brain for any reason (cancerous or non-cancerous tumors, subdural hematomas, AV malformations, increased intracranial pressure, etc.)
* Participant report of a history of stroke (with the exception of TIA if ≥1 year ago)
* Participant report of HIV/AIDS
* Participant report of moderate to severe head trauma (loss of consciousness > 60 min or with evidence of structural brain changes on imaging)
* History of major psychiatric disorder (DSM-IV Axis 1) (i.e. major depressive disorder (untreated or poorly treated), bipolar disorders, schizophrenia, or substance abuse disorders (self-reported and/or stated in medical record).
* Participant report of a history of prior breast or other cancer with the exception of non-melanoma skin cancer. An exception for cases only: women who completed treatment for a previous cancer at least 5 years ago and have not undergone any chemotherapy or hormonal therapy. This previous cancer cannot be breast cancer.
* Participant report of previous or current chemotherapy or hormonal therapy use
* Participant use of methotrexate (Amethopterin, Rhematrex, Trexall) or rituximab (Rituxin) for rheumatoid arthritis, psoriasis or Crohn's disease, or cyclophosphamide (Cytoxan, Neosar) for Lupus.
* Visual or hearing impairment that would preclude ability to complete interviews or neuropsychological testing, such as significant macular degeneration or being unable to correct hearing with hearing aides
* Non-English speaking
* To participate in the optional neuroimaging portion of the study:

Participant cannot be claustrophobic Participant cannot have a pacemaker, aneurysm clip or other implants that are not MRI safe Participant cannot have any type of implanted electrical device

Ages: 60 Years to 105 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female breast cancer cases and female matched non-cancer controls
Study Population: Women age 60+ with a newly diagnosed breast adenocarcinoma staged 0-3 and matched controls.
Sampling Method: Non-Probability Sample
Enrollment: 1700 (Estimated)
Dates: Start 2010-08-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Attention, Processing Speed, Executive Function (APE) Domain | Baseline and annually up to 5 years
  Using neuropsychological tests: NAB Digits Forward and Backward, Trailmaking A and B, Digit Symbol Subtest-Wechsler Adult, The Timed Instrumental Activities of Daily Living, Controlled Oral Word Association Test, NAB Driving Scenes and NAB Figure Drawing. These measures are aggregated to arrive at one reported value. The individual tests are first selected via factor analysis, then the selected raw scores are standardized to baseline controls by age and education group. The final domain score is calculated by averaging available individual z-standardized test scores.
Change in Learning and Memory (LM) Domain | Baseline and annually up to 5 years
  Using neuropsychological tests: Logical Memory I and II (Wechsler Memory Scale), NAB List Learning (Immediate Recall, Short Delay Recall, Long Delay). These measures are aggregated to arrive at one reported value. The individual tests are first selected via factor analysis, then the selected raw scores are standardized to baseline controls by age and education group. The final domain score is calculated by averaging available individual z-standardized test scores.
Change in Cognition Domain | Baseline and annually up to 5 years
  Using assessment: FACT-Cog and PCI Sub-scale. The measures are aggregated to arrive at one reported value. Change in cognition is calculated based on the official FACT-Cog scoring manual.
  The total score is calculated by summing the available items among all 37 items when no more than 30 items are missing.
  The PCI subscale score is calculated by summing the available items among all 18 items when no more than 8 items are missing.

SECONDARY OUTCOMES:
Change in Quality of Life | Baseline and annually up to 5 years
  Using Functional Assessment of Cancer Therapy-Breast quality of life measure (FACT-B)
Change in Quality of Life | Baseline and annually up to 5 years
  Using Medical Outcome Study measure (MOS)
Change in Quality of Life | Baseline and annually up to 5 years
  Using Short Form Health Survey measure (SF-12)
Change in cancer-related symptoms (including fatigue, sleep, pain, anxiety and depression) | Baseline and annually up to 5 years
  Using survey data
Biomarkers of aging (genotype, inflammatory biomarkers, telomere length, p16, miRNA) | Baseline and annually up to 5 years
  Using annual biospecimen collection of blood or saliva
Grip Strength Test | Baseline and annually up to 5 years
  Participant's grip strength will be measured using the Jamar Plus Digital dynamometer. The participant should be in a standing position, arms at their side, not touching their body with elbow bent slightly. If subjects are unable to stand comfortably, they will be seated in a chair with their feet touching the ground with their elbow bent to 90 degrees and the arm against their trunk with a neutral wrist. Participants squeeze the Jamar Plus Digital dynamometer as hard as they can for a count of three. The dynamometer provides a digital reading of force in pounds. A practice trial at less than full force and one test trial are completed with each hand. The test takes approximately three minutes to administer. Dominant vs. Non-Dominant Hand (i.e., handedness) is assessed at the outset.
Actigraphy/Change in Sleep | Baseline and annually up to 5 years
  To obtain an objective assessment of both daytime and nighttime sleeping, participants will wear the actigraph on the dominant wrist (unless that arm is paralyzed) for one week. The Actigraph Motionlogger (Ambulatory Monitoring, Inc. Ardsley, NY), is a wrist-mounted actigraph that records activity and illumination exposure using an accelerometer, a light transducer and a microprocessor. Commercially available software uses validated algorithms that take into account wrist movement immediately before and after an epoch of interest; wrist activity below an established threshold is interpreted as sleep and wrist activity above that threshold is interpreted as wakefulness as validated in older adults. Agreement between wrist actigraphy and EEG (the gold standard method for sleep assessment) scoring of sleep variables (e.g., total sleep time) is 89-95% in older adults.

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne Mandelblatt, Principal Investigator — Lombardi Comprehensive Cancer Center
Locations (1):
- Georgetown University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McDonald BC, Van Dyk K, Deardorff RL, Bailey JN, Zhai W, Carroll JE, Root JC, Ahles TA, Mandelblatt JS, Saykin AJ. Multimodal MRI examination of structural and functional brain changes in older women with breast cancer in the first year of antiestrogen hormonal therapy. Breast Cancer Res Treat. 2022 Jul;194(1):113-126. doi: 10.1007/s10549-022-06597-1. Epub 2022 Apr 27. PMID 35476252
- [Derived] Bethea TN, Zhai W, Zhou X, Ahles TA, Ahn J, Cohen HJ, Dilawari AA, Graham DMA, Jim HSL, McDonald BC, Nakamura ZM, Patel SK, Rentscher KE, Root J, Saykin AJ, Small BJ, Van Dyk KM, Mandelblatt JS, Carroll JE. Associations between longitudinal changes in sleep disturbance and depressive and anxiety symptoms during the COVID-19 virus pandemic among older women with and without breast cancer in the thinking and living with breast cancer study. Cancer Med. 2022 Sep;11(17):3352-3363. doi: 10.1002/cam4.4682. Epub 2022 Mar 22. PMID 35315588
- [Derived] Dilawari A, Rentscher KE, Zhai W, Zhou X, Ahles TA, Ahn J, Bethea TN, Carroll JE, Cohen HJ, Graham DA, Jim HSL, McDonald B, Nakamura ZM, Patel SK, Root JC, Small BJ, Saykin AJ, Tometich D, Van Dyk K, Mandelblatt JS; Thinking and Living with Cancer Study. Medical care disruptions during the first six months of the COVID-19 pandemic: the experience of older breast cancer survivors. Breast Cancer Res Treat. 2021 Nov;190(2):287-293. doi: 10.1007/s10549-021-06362-w. Epub 2021 Sep 13. PMID 34515905
- [Derived] Carroll JE, Small BJ, Tometich DB, Zhai W, Zhou X, Luta G, Ahles TA, Saykin AJ, Nudelman KNH, Clapp JD, Jim HS, Jacobsen PB, Hurria A, Graham D, McDonald BC, Denduluri N, Extermann M, Isaacs C, Dilawari AA, Root J, Stern RA, Mandelblatt JS; Thinking and Living With Cancer Study. Sleep disturbance and neurocognitive outcomes in older patients with breast cancer: Interaction with genotype. Cancer. 2019 Dec 15;125(24):4516-4524. doi: 10.1002/cncr.32489. Epub 2019 Sep 25. PMID 31553501
- [Derived] Tometich DB, Small BJ, Carroll JE, Zhai W, Luta G, Zhou X, Kobayashi LC, Ahles T, Saykin AJ, Clapp JD, Jim HSL, Jacobsen PB, Hurria A, Graham D, McDonald BC, Denduluri N, Extermann M, Isaacs C, Dilawari A, Root J, Rini C, Mandelblatt JS; Thinking and Living with Cancer (TLC) Study. Pretreatment Psychoneurological Symptoms and Their Association With Longitudinal Cognitive Function and Quality of Life in Older Breast Cancer Survivors. J Pain Symptom Manage. 2019 Mar;57(3):596-606. doi: 10.1016/j.jpainsymman.2018.11.015. Epub 2018 Nov 23. PMID 30472317

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-09): https://cdn.clinicaltrials.gov/large-docs/83/NCT03451383/Prot_SAP_003.pdf